CLINICAL TRIAL: NCT04834661
Title: Safety and Feasibility of Performing Laparoscopic Surgery for Colorectal and Gastric Cancer Outside the Primary Registered Medical Institution Under Multi-sites Practice (MSP) Policy, a Retrospective Comparative Study
Brief Title: Performing Laparoscopic Surgery for Colorectal and Gastric Cancer Outside the Primary Registered Medical Institution
Status: Completed | Type: Observational
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Principal Investigator, Cai Zhenghao, Attending surgeon of gastrointestinal surgery，Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai Minimally Invasive Surgery Center
Other Study IDs: multi-sites practice surgery
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Colorectal Cancer; Gastric Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- inside group: laparoscopic surgery for colorectal and gastric cancer inside the primary registered medical institution
  Interventions: Other: surgery inside the primary institution
- outside group: laparoscopic surgery for colorectal and gastric cancer outside the primary registered medical institution
  Interventions: Other: surgery outside the primary institution

INTERVENTIONS:
Other: surgery inside the primary institution — to perform laparoscopic surgery for colorectal and gastric cancer inside the primary registered medical institution
  Groups: inside group
Other: surgery outside the primary institution — to perform laparoscopic surgery for colorectal and gastric cancer outside the primary registered medical institution
  Groups: outside group

SUMMARY:
This study investigates the safety and feasibility of performing laparoscopic surgery for colorectal and gastric cancer inside versus outside the primary registered medical institution under multi-sites practice (MSP) policy. This is a single practitioner, retrospective comparative study. The endpoints are peri-operative outcomes, pathological results, and medical costs.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 100 years
* diagnosed as colorectal cancer or gastric cancer
* undergoing laparoscopic surgery between 2016-2020 performed by Dr Feng

Exclusion Criteria:

* Emergency procedure
* without histopathological result of malignancy
* conventional open surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: colorectal cancer and gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 1130 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
overall postoperative complication rate | 30 days after surgery
  postoperative complications evaluated according to Clavin-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Zhenghao Cai, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China